CLINICAL TRIAL: NCT00156208
Title: A Phase III, 18-Month, Extension Study to Evaluate the Safety of Asoprisnil in Subjects With Uterine Leiomyomata
Brief Title: Safety of Treatment of Uterine Fibroids With Asoprisnil
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Cynthia Mattia-Goldberg, Abbott
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C03-062
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2008-05

CONDITIONS: Fibroid Uterus; Leiomyoma; Menorrhagia; Metrorrhagia; Uterine Fibroids
Keywords: Symptomatic Uterine Fibroids; Excessive Uterine Bleeding; Uterine Hemorrhage; asoprisnil
MeSH Terms: conditions — Leiomyoma; Menorrhagia; Metrorrhagia; Uterine Hemorrhage | interventions — asoprisnil

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Asoprisnil
- 2 (Experimental)
  Interventions: Drug: Asoprisnil

INTERVENTIONS:
Drug: Asoprisnil — 10mg Tablet, oral Daily for 18 months
  Other Names: J867
  Arms: 1
Drug: Asoprisnil — 25 mg Tablet, oral Daily for 18 months
  Other Names: J867
  Arms: 2

SUMMARY:
The objective of this study is to determine the long-term safety of asoprisnil in women with symptomatic uterine fibroids who completed the 6 month Study C02-037.

DETAILED DESCRIPTION:
No medical therapy is currently available for the long-term treatment of abnormal uterine bleeding associated with uterine fibroids in women and many women must resort to surgery for relief. The objective of this study is to determine the long-term safety of asoprisnil 10 and 25 mg administered daily for 18 months to subjects with symptomatic uterine leiomyomata who completed the 6 month Study C02-037. The safety endpoints for this study will be based on assessments of the endometrium, ovarian cysts, lipid profiles, adverse events and clinical laboratory evaluations.

Some subjects receiving asoprisnil developed endometrial changes. As a result, dosing was prematurely discontinued for all subjects. To ensure safety, subjects will remain on study and will undergo scheduled study procedures. In most subjects, endometrial changes reversed after asoprisnil discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Women that have completed 6 months of treatment in study C02-037 with no more than a 7-day interruption in their treatment
* Otherwise good health
* Premenopausal based on Estrogen and Follicle Stimulating Hormone levels
* Agrees to double-barrier method of contraception
* Adequate endometrial biopsy with no significant histological disorder

Exclusion Criteria:

* Any abnormal lab or procedure result(s) the study-doctor considers important
* History of a blood-clotting disorder
* Any prior surgical and/or invasive procedure(s) for uterine fibroids that resulted in either a cure or made the symptoms go away
* Significant gynecological disorder, such as endometrial polyp

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2004-04; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Long Term Safety | Throughout 18 month treatment period

SECONDARY OUTCOMES:
Cumulative and incremental amenorrhea rates. | Each month 1-18
Change from baseline in total symptom severity score and the Uterine Fibroid Symptoms-Quality of Life total score. | Final Visit
Change from baseline in menorrhagia, metrorrhagia, bloating, pelvic pressure, dysmenorrhea, pelvic pain and urinary symptoms. | Final Visit
Change from baseline in Uterine Fibroid Impact Questionnaire. | Months 6, 12, 18
Change from baseline in the Work Limitation Questionnaire Index. | Final Visit
Change from baseline in the two dimensions of the SF-36. | Final Visit
Change from baseline in the monthly bleeding score. | Final Month
Change from baseline in the hemoglobin concentration. | Final Visit
Percent change from baseline in volume of the largest fibroid. | Final Visit
Percentage of subjects who discontinue with the intent to have surgery for fibroids. | During Treatment Period
Percentage of subjects who responded positively to the Global Efficacy Questions. | Months 6, 12, 18

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Chair — Abbott